CLINICAL TRIAL: NCT00104169
Title: Pilot Study of Epoetin Alfa in Idiopathic Anemia of Aging (IAA)
Brief Title: Idiopathic Anemia of Aging (IAA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No subject accrual
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: AG0014
Record Dates: First submitted 2005-02-23; First posted 2005-02-24 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Anemia; Aging
Keywords: Anemia; Frailty; Epoetin; Erythropoietin; EPO
MeSH Terms: conditions — Anemia; Frailty | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin Alfa

SUMMARY:
The purpose of this trial is to examine whether Epoetin Alfa, a hormone stimulating production of red blood cells, can reverse idiopathic anemia.

DETAILED DESCRIPTION:
As individuals become older, the frequency of anemia increases. While the cause of anemia in many cases can be determined and corrected, in a number of individuals there is no correctable cause found and the patient must live with their anemia. This is known as idiopathic anemia, and can have serious consequences for the individual. Numerous studies have demonstrated that anemia is associated with loss of energy and stamina, causing individuals to decrease their activities, which adversely affects both their sense of well-being as well as their physical strength. Losses in these areas are associated with the clinical manifestations of frailty.

The current pilot study will examine whether or not administration of Epoetin Alfa, a hormone stimulating production of red blood cells, can reverse this type of anemia. We will examine the consequences of reversing the anemia in terms of physical strength and function, cardiovascular function and sense of well-being and mental function.

In this study, individuals with anemia will be treated for six months with Epoetin Alfa following the correction of their anemia and measurements done to evaluate physical strength, performance, cardiac, mental and kidney function. At the end of treatment, individuals will be followed for an additional six months to determine whether the anemia recurs and physical function decreases.

Participation in this study is voluntary. All testing and medication received are free to the participant.

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age or older
* Diagnosed with anemia
* Hemoglobin level less than or equal to 11
* Able to perform most activities of daily living without restriction

Exclusion Criteria:

* History of serious heart, liver or kidney disease
* Cancer treated within the last year except for skin cancer (excluding melanoma)
* Problems with your immune system
* Received Epoetin Alfa within the last year

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Response of Anemia

SECONDARY OUTCOMES:
To determine if there is a beneficial effect of quality of life, cognitive function, and physical function.

CONTACTS AND LOCATIONS:
Overall Officials: William Ershler, MD, Principal Investigator — NIA, NIH
Locations (1):
- Harbor Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Cesari M, Penninx BW, Lauretani F, Russo CR, Carter C, Bandinelli S, Atkinson H, Onder G, Pahor M, Ferrucci L. Hemoglobin levels and skeletal muscle: results from the InCHIANTI study. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):249-54. doi: 10.1093/gerona/59.3.m249. PMID 15031309
- [Background] Guralnik JM, Eisenstaedt RS, Ferrucci L, Klein HG, Woodman RC. Prevalence of anemia in persons 65 years and older in the United States: evidence for a high rate of unexplained anemia. Blood. 2004 Oct 15;104(8):2263-8. doi: 10.1182/blood-2004-05-1812. Epub 2004 Jul 6. PMID 15238427
- [Background] Penninx BW, Guralnik JM, Onder G, Ferrucci L, Wallace RB, Pahor M. Anemia and decline in physical performance among older persons. Am J Med. 2003 Aug 1;115(2):104-10. doi: 10.1016/s0002-9343(03)00263-8. PMID 12893395
- [Background] Chaves PH, Ashar B, Guralnik JM, Fried LP. Looking at the relationship between hemoglobin concentration and prevalent mobility difficulty in older women. Should the criteria currently used to define anemia in older people be reevaluated? J Am Geriatr Soc. 2002 Jul;50(7):1257-64. doi: 10.1046/j.1532-5415.2002.50313.x. PMID 12133021
- [Background] Kikuchi M, Inagaki T, Shinagawa N. Five-year survival of older people with anemia: variation with hemoglobin concentration. J Am Geriatr Soc. 2001 Sep;49(9):1226-8. doi: 10.1046/j.1532-5415.2001.49241.x. PMID 11559383